CLINICAL TRIAL: NCT03939650
Title: Differential Diagnosis Assessment in Ambulatory Care With an Automated Medical History-Taking Device: A Confirmatory Pseudo-Randomized Study With Accurate Gold-standard Diagnosis
Brief Title: Diagnosis Assessment With Diaana #3
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: logistics: not able to get resosurces to beginn
Sponsor: Adrien Schwitzguebel (Other)
Responsible Party: Sponsor-Investigator, Adrien Schwitzguebel, Medical doctor & principal investigator, Hôpital de la Providence, Switzerland
Organization: Hôpital de la Providence, Switzerland (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: COLLINE_Diaana
Record Dates: First submitted 2019-05-03; First posted 2019-05-07 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2019-10

CONDITIONS: Decision Making; Computer-assisted; General Practitioners; Patient Engagement
Keywords: differential diagnosis; hospital outpatient clinics; clinical applications software
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Intervention Model Description: For each of the six resident physicians of the outpatients clinic, the 6 first eligible patients will be attributed to the control group (with access to "Diaana"), then the 12 next eligible patients will be attributed to the interventional group (with access to "Diaana"). There will therefore be 36 patients in the control group and 72 in the interventional group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaana (Experimental): 1. The patient fulfill Diaana
  2. The resident physician reads the Diaana summary
  3. The resident physician see the patient in consultation. He establishes his DD without having access to the complementray exams (blood tests, x-ray, ...)
  4. The senior physician see the patient at the follow-up consultation. He establishes the gold-standard diagnosis highlighted by complementary exams and imagery.
  Interventions: Device: Diaana
- Control (No Intervention): 1. The resident physician see the patient in consultation. He establishes his DD without having access to the complementray exams (blood tests, x-ray, ...)
  2. The senior physician see the patient at the follow-up consultation. He establishes the gold-standard diagnosis highlighted by complementary exams and imagery.

INTERVENTIONS:
Device: Diaana — Diaana, the AMHTD used, functions as follows: on the basis of an interactive questionnaire completed by the patient before the consultation, it performs an exhaustive anamnesis focused on the problem and proposes a panel of DDs with a high sensitivity. The artificial reasoning system of "Diaana" mimics how a specialist physician would reason to establish a DD. The information transmitted is in an easy-to-use form for the physician that includes a summary of the anamnesis centered on relevant elements from the questionnaire and a list of possible diagnoses with their emergency level, potential contributing factors, and first-line management proposals.
  Other Names: Automated medical history-taking device (AMHTD)
  Arms: Diaana

SUMMARY:
Single-center, unblinded, 2:1 parallel pseudo-randomized efficacy trial.

In the intervention group only, resident physicians will be assisted by the automated medical history-taking device "Diaana" during their consultations in outpatient ambulatory unit of the Geneva University Hospital.

In both groups, the differential diagnosis of the resident physician will be compared to the gold-standard diagnosis of the senior physician.

DETAILED DESCRIPTION:
Automated medical history-taking devices (AMHTD) are emerging tools with the potential to increase the quality of medical consultations by providing physicians with an exhaustive, high-quality, standardized anamnesis and differential diagnosis. In this study, the investigators aimed to establish whether an AMHTD of interest, "Diaana", allowed the physician to establish a more precise differential diagnosis.

A single-center, unblinded, 2:1 parallel pseudo-randomized efficacy trial will be performed. A consultation follow-up is organized at 4-6 weeks, were the gold-standard diagnosis is established by the senior physician. The study will take place in the emergency outpatient unit of La Colline Hospital (Geneva, Switzerland) and include patients suffering from symptoms covered by Diaana.

Patients in the intervention group will fulfill Dianna. Then, the resident physician will read Diaana summary, perform his consultation, and fulfill case report form, including his differential diagnosis. Then, the senior physician will see the patient and establish the gold-standard diagnosis. In the control group, the residents will directly establish a differential diagnosis, without the help of Diaana.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the emergency outpatient unit of La Colline hospital (Geneva, Switzerland)
* Patients suffering from symptoms localized to the superior or inferior member, the back, hand the chest wall.

Exclusion Criteria:

* Strictly dermatologic concerns
* Toes trauma (because the diagnosis of those conditions is generally obvious)
* Medical condition considered as urgent
* Inability to complete de digilatized Diaana form (sight problems, language, inability to use a tablet computer)

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-31 (Estimated); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the diagnosis established by the resident physician | At day 0
  The resident physician will select up to 5 diagnose in an exhaustive list, from the most to the least relevant.
  The accuracy of the diagnosis established will be measured as following:
  * 100% if the gold-standard diagnosis is in position#1 into the resident diagnosis list
  * 80% if the gond-standard diagnosis is in position#2
  * 60% in position #3
  * 40% in position #4
  * 20% in position #5
  * 0% if the gold-standard diagnosis absent of the resident diagnosis list
  A higher percentage is considered as a better outcome.

SECONDARY OUTCOMES:
Consultation time | At day 0
  The resident's consultation (with and without the patient) will be measured by the research coordinator. Consultation time will be compared between groups. A shorter consultation time will be considered as a better outcome.
Patient satisfaction: Likert 1-4 scale | At day 0
  Into the experimental group, the patient's satisfaction will be evalatued on a Likert 1-4 scale. 1= fully dissatisfied; 2 = partially dissatisfied; 3 = partially satisfied; 4 = fully satisfied A higher score is considered as a better outcome.
Differential diagnosis established by Diaana | At day 0
  The Diaana system will select diagnoses in an exhaustive list. The percentage of cases were the gold-standard diagnosis is present into the differential diagnosis list will be measured. A higher percentage is a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- La Colline Hospital Outpatient Unit, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No